CLINICAL TRIAL: NCT06140407
Title: A Single Arm Trial of Adjuvant Pembrolizumab in Patients With Limited Stage Small Cell Lung Cancer
Brief Title: Pembrolizumab After Radiation Therapy and Chemotherapy in Limited Stage Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual and Merck discontinuing funding and drug supply
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Ryan Whitaker, Assistant Professor of Medicine, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICCTHO22114; NCI-2023-09018 (Registry Identifier: NCI, Clinical Trials Reporting Program)
Record Dates: First submitted 2023-11-01; First posted 2023-11-20 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Limited Stage Lung Small Cell Carcinoma; Stage I Lung Cancer; Stage II Lung Cancer; Stage III Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Cisplatin; Carboplatin; Etoposide; pembrolizumab; Magnetic Resonance Spectroscopy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pembrolizumab) (Experimental): Patients undergo radiation therapy and receive cisplatin or carboplatin on day 1 of each cycle and etoposide on days 1-3 for 4 cycles. Patients then receive pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days for 1 year in the absence of disease progression or unacceptable toxicity. Patients undergo PET scan during screening. Patients also undergo MRI throughout the trial as well as CT. Additionally, patients undergo blood sample collection throughout the trial.
  Interventions: Drug: Cisplatin; Drug: Carboplatin; Drug: Etoposide; Biological: Pembrolizumab; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Biospecimen Collection; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Cisplatin — Receive Cisplatin
Drug: Carboplatin — Receive Carboplatin
Drug: Etoposide — Receive Etoposide
Biological: Pembrolizumab — Receive Pembrolizumab by IV
Procedure: Computed Tomography — Undergo Computed Tomography
Procedure: Positron Emission Tomography — Undergo Positron Emission Tomography
Procedure: Magnetic Resonance Imaging — Undergo Magnetic Resonance Imaging
Procedure: Biospecimen Collection — Undergo blood sample collection
Radiation: Radiation Therapy — Undergo Radiation Therapy

SUMMARY:
This phase II trial studies how well pembrolizumab after standard treatment with radiation plus the following chemotherapy drugs: cisplatin or carboplatin, plus etoposide works in treating patients with limited stage small cell lung cancer (LS-SCLC). Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving pembrolizumab after standard treatment with radiation plus chemotherapy may increase the ability of the immune system to fight LS-SCLC.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To investigate progression free survival per Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) as assessed by the investigator in patients with limited stage small cell lung cancer treated with adjuvant pembrolizumab.

SECONDARY OBJECTIVES:

I. Assess median overall survival compared to the historical control dataset (CONVERT trial1) median overall survival (OS) of 30 months.

II. Assess the safety and tolerability of adjuvant pembrolizumab in patients with limited stage SCLC.

EXPLORATORY/TRANSLATIONAL OBJECTIVES:

I. To determine whether patients with detectable circulating tumor deoxyribonucleic acid (ctDNA) after curative intent therapy ("minimal residual disease [MRD] positive") experience shorter median progression free survival (PFS) compared to patients without detectable ctDNA after curative intent therapy ("MRD negative.").

II. Determination of whether patients with ctDNA clearance at any point during curative intent therapy have superior median PFS compared to patients who do not experience ctDNA clearance during curative intent therapy.

OUTLINE:

Patients undergo radiation therapy and receive cisplatin or carboplatin on day 1 of each cycle and etoposide on days 1-3 for 4 cycles. Patients then receive pembrolizumab intravenously (IV) over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days for 1 year in the absence of disease progression or unacceptable toxicity. Patients undergo positron emission tomography (PET) scan during screening. Patients also undergo magnetic resonance imaging (MRI) throughout the trial as well as computed tomography (CT). Additionally, patients undergo blood sample collection throughout the trial.

After completion of study treatment, patients are followed up at 30 days, and every 12 weeks for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Has LS-SCLC (stage I-III, by American Joint Committee on Cancer [AJCC] 8th Edition Cancer Staging) and no evidence of extensive stage disease. Participants may enroll at any time between diagnosis and initiation of definitive concurrent chemoradiation or surgery followed by adjuvant chemotherapy. Correlative analyses collected during standard of care definitive concurrent chemoradiation or surgery followed by adjuvant chemotherapy are mandatory
* Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of small cell lung cancer or high grade neuroendocrine carcinoma will be enrolled in this study
* Contraception requirements should conform with Clinical Trials Facilitation and Coordination Group (CTFG) guidelines. The pembrolizumab standard for use of highly effective contraceptive methods for persons of child-bearing potential (POCBP) is 120 days (5 half-lives) after the last dose. Please either list the contraception requirement for each compound in the study or use the longest time frame that covers requirements for all compounds in the study
* Similarly, Company standard for abstaining from breastfeeding after study intervention is at least 5 half-lives. For pembrolizumab, this is 120 days
* No radiological imaging evidence of disease progression after completion of definitive concurrent chemoradiation or surgery followed by adjuvant chemotherapy
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention
* Participants who are hepatitis B surface antibody (HBsAg) positive are eligible if they have received hepatitis B virus (HBV) anti-viral therapy for at least 4 weeks, and have undetectable HBV viral load prior to randomization.

Note: Participants should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention.

Hepatitis B screening tests are not required unless:

* Known history of HBV infection
* As mandated by local health authority

  • Participants with a history of hepatitis C virus (HCV) infection are eligible if HCV viral load is undetectable at screening. Hepatitis C screening tests are not required unless:
* Known history of HCV infection
* As mandated by local health authority Note: Participants must have completed curative anti-viral therapy at least 4 weeks prior to randomization

  • Human immunodeficiency virus (HIV)-infected participants must have well-controlled HIV on antiretroviral therapy (ART), defined as:
* Participants on ART must have a CD4+ T-cell count >= 350 cells/mm^3 at the time of screening
* Participants on ART must have achieved and maintained virologic suppression defined as confirmed HIV ribonucleic acid (RNA) level below 50 or the lower limit of quantitation (LLOQ) (below the limit of detection) using the locally available assay at the time of screening and for at least 12 weeks before screening
* It is advised that participants must not have had any acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections within the past 12 months.
* Participants on ART must have been on a stable regimen, without changes in drugs or dose modification, for at least 4 weeks before study entry (day 1) and agree to continue ART throughout the study
* The combination ART regimen must not contain any antiretroviral medications that interact with CYP3A4 inhibitors/inducers/substrates (https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-and-drug-interactions-table-substrates-inhibitors-and-inducers)

  * Absolute neutrophil count (ANC) >= 1500/uL (specimens must be collected within 10 days prior to the start of study intervention)
  * Platelets >= 100000/uL (specimens must be collected within 10 days prior to the start of study intervention)
  * Hemoglobin ≥ 9.0 g/dL or ≥ 5.6 mmol/L (specimens must be collected within 10 days prior to the start of study intervention)
* Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks

  • Creatinine or measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine Clearance [CrCl]) =< 1.5 X upper limit of normal (ULN) or >= 30 mL/min for participant with creatinine levels > 1.5 X institutional ULN (specimens must be collected within 10 days prior to the start of study intervention)
* Creatinine clearance (CrCl) should be calculated per institutional standard

  * Total bilirubin =< 1.5 X ULN or direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 X ULN (specimens must be collected within 10 days prior to the start of study intervention)
  * Alanine aminotransferase (AST) (serum glutamic pyruvic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 X ULN (specimens must be collected within 10 days prior to the start of study intervention)
  * International normalized ratio (INR) or prothrombin time (PT) activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants (specimens must be collected within 10 days prior to the start of study intervention)

Exclusion Criteria:

* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137)
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to allocation
* Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities requiring corticosteroids, and not have had radiation pneumonitis. The last radiotherapy treatment must have been performed at least 7 days before the first dose of study drug
* Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of pembrolizumab
* Has a known additional malignancy that is progressing or requires active treatment. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, localized prostate adenocarcinoma, or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded. Participants with low-risk early-stage prostate cancer (T1-T2a, Gleason score =< 6, and prostate-specific antigen [PSA]< 10 ng/mL) untreated in active surveillance with stable disease are not excluded
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has severe hypersensitivity (≥ grade 3) to pembrolizumab
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has an active infection requiring systemic therapy
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment
* Has had an allogenic tissue/solid organ transplant
* Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* HIV-infected participants with a history of Kaposi's sarcoma and/or Multicentric Castleman's Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-02-14 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Time from the date of first treatment to progressive disease or death due to any cause, whichever occurs first, assessed up to 3 years

SECONDARY OUTCOMES:
Overall survival | Time from the date of first treatment to the date of death due to any cause, assessed up to 3 years
Incidence of adverse events | Up to 3 years
  Will be assessed by National Cancer Institute's Common Terminology Criteria for Adverse Events version 5.0. Toxicities will be characterized in terms regarding seriousness, causality, toxicity grading, and action taken with regard to trial treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Whitaker, MD, PhD, Principal Investigator — Vanderbilt University/Ingram Cancer Center
Locations (1):
- Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2024-05-03): https://cdn.clinicaltrials.gov/large-docs/07/NCT06140407/ICF_000.pdf